CLINICAL TRIAL: NCT01976143
Title: A Phase 1 Study to Evaluate the Effect of Nktr-102 for Injection (Etirinotecan Pegol) on the QT/QTC Interval in Patients With Advanced or Metastatic Solid Tumors
Brief Title: A Study in Cancer Patients to Evaluate the Effect of a Single Dose of NKTR-102 (Etirinotecan Pegol) on the QTc Interval and to Assess Pharmacokinetics and Safety
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nektar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-102-12
Record Dates: First submitted 2013-10-29; First posted 2013-11-05 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Advanced Cancer; Metastatic Solid Tumors
MeSH Terms: interventions — etirinotecan pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NKTR-102 (Experimental): A single 90 minute IV infusion of 220 mg/m2 NKTR-102
  Interventions: Drug: NKTR-102

INTERVENTIONS:
Drug: NKTR-102

SUMMARY:
The purpose of this research study is to evaluate the effect of NKTR-102 on the QT/QTc interval in patients with advanced or metastatic solid tumors

DETAILED DESCRIPTION:
This is an open-label study that will assess the effect of NKTR- 102 on cardiac ventricular repolarization, as characterized by QTcF (QT interval with Fridericia correction) interval values, in patients with advanced or metastatic solid tumors following administration of a single dose of NKTR-102.

ELIGIBILITY:
Inclusion Criteria:

* Advanced or metastatic solid tumor refractory to standard therapy
* Measurable or non-measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Resolution of acute toxic effects of prior chemotherapy and other cancer treatments
* Left ventricular ejection fraction (LVEF) ≥50% by echocardiogram
* Adequate bone morrow and organ function
* Electrolytes within normal limits
* Stopped tobacco use for 4 weeks prior to day 1 and during the study
* Agree to use adequate contraception

Exclusion Criteria:

* Previous anti-cancer therapy for malignancy within 4 weeks (6 weeks for the nitrosoureas or mitomycin C) before day 1
* Treatment with antiarrythmic drugs and any medication known to cause QTc prolongation within 4 weeks before screening and during the study
* Prior extensive anthracycline exposure
* Administration of cytochrome P450 CYP3A4 inducers and inhibitors within 4 weeks before day 1 and during the study
* Intake of grapefruit, grapefruit juice, Seville oranges, or other products containing grapefruit or Seville oranges within 14 days prior to day 1 and during the study
* History of serious cardiovascular disease
* Abnormal systolic blood pressure, diastolic blood pressure and/or heart rate
* History of additional risk factors for Torsade de Pointes
* Prolonged QTcF
* Important abnormalities of the ECG that may interfere with the interpretation of QTc interval changes at screening
* Implantable pacemaker or automatic implantable cardioverter defibrillator
* UGT1A1 genotype of TA 7 in both alleles (homozygous UGT1A1*28) or TA 8 in either one or both alleles (hetero- or homozygous for UGT1A1*37)
* Any major surgery within 4 weeks prior to day 1
* Concurrent treatment with other anticancer therapy
* Untreated central nervous system metastases
* Chronic or acute GI disorders resulting in diarrhea
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-02; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
QTcF interval values | Day -1 through Day 42
  10 pre-dose and 18 post-dose ECG measurements to evaluate the effect of NKTR-102

SECONDARY OUTCOMES:
Pharmacokinetics (PK) and ECG Parameters | Day 1 through Day 42
  1 pre-dose and 18 post-dose blood samples to measure concentrations of NKTR-102 and its metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Gergel, MD, Study Director — Nektar Therapeutics
Locations (3):
- United States (3):
  - American Institute of Research, Los Angeles, Los Angeles, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University Hospitals Case-Medical Center Seidman Cancer Center, Cleveland, Ohio